CLINICAL TRIAL: NCT02350088
Title: Fast-track Surgery in the Treatment of Hirschsprung's Disease
Acronym: Fast-track
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jiexiong Feng, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tongji Fast-track surgery
Record Dates: First submitted 2015-01-17; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Surgery
Keywords: fast-track surgery
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fast-track Surgery (Active Comparator): probiotics,oral,b.i.d.
  Interventions: Drug: probiotics
- Traditional Group (Active Comparator): placebo,oral,b.i.d.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: probiotics — probiotics
  Other Names: Bifico
  Arms: Fast-track Surgery
Drug: placebo — placebo
  Other Names: Bifico
  Arms: Traditional Group

SUMMARY:
To evaluate the safety and efficacy of Hirschsprung's disease

DETAILED DESCRIPTION:
The patients are divided into two groups：fast-track surgery combined with laparoscope group and laparoscope with traditional managements group.Postoperative recovery,hospital stay,hospital cost and complcations were compared.

ELIGIBILITY:
Inclusion Criteria:

1. surgical treatment for Hirschsprung's disease
2. The first procedure for Hirschsprung's disease
3. Age<14 years

Exclusion Criteria:

1. conservative treatment for Hirschsprung's disease
2. The reoperation for Hirschsprung's disease
3. Age>14 years

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
number of participants with recovery of boewl movements | one year

SECONDARY OUTCOMES:
Duration of the hospital stay | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Li, MD PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China